CLINICAL TRIAL: NCT01814254
Title: Comparison of Body Hydration State in Hemodialysis Patients With the Hydra 4200 and ZOE (100 and 5 kHZ) Bioimpedance Devices
Brief Title: Comparison of Body Hydration State in Hemodialysis Patients
Status: Terminated | Type: Observational
Why Stopped: Change of Institutional Affiliation & Funding
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 063-11
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Hemodialysis; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Receiving hemodialysis

SUMMARY:
Estimation of hydration state in dialysis patients is a major challenge in clinical practice. Although many methods have been studied, none have been established yet for clinical routine practice.

The investigators have developed a method, using segmental and calf bioimpedance spectroscopy (cBIS) techniques to measure body hydration. The device we used based on the FDA-approved Hydra 4200 (Xitron Technologies, San Diego, CA). The Hydra 4200 was initially developed to measure whole body and segmental body fluid volumes but Hydra is approved only for measuring healthy subjects. The cBIS monitors hydration state by continuously measuring change in resistance and resistivity in the calf during hemodialysis (HD) or it can be used for simple measurement before, during and after dialysis. Preliminary results in clinical studies have shown that optimal hydration state of HD patients may be determined by the calf method. This study aims to compare the Hydra 4200 to two other devices: the FDA approved ZOE (100 kHz) Fluid Status Monitor (Noninvasive Medical Technologies, Inc, Las Vegas) and a modified version ZOE 5 kHz. The modified ZOE monitor (ZOE (5 kHz)) delivers frequency of 5 kHz and 0.8 mA current instead of 100 kHz and 2 mA.

The subjects of this study include a group of hemodialysis patients and a group of healthy controls. The healthy controls are used to identify a normal range within the healthy population for each method. Each hemodialysis patient will be studied twice in different hydration state. The study will not change the procedure of the patient's dialysis treatment. Since all devices are based on noninvasive bioimpedance technique, this study has minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable

Exclusion Criteria:

* Implants including pacemakers, implantable pumps, artificial joints
* Limb amputations
* Pregnancy
* Simultaneous participation in another clinical study except observational trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis clinics
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Calf bioimpedance measurement | 2 dialysis treatments within 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Yorkville Dialysis, New York, New York, United States